CLINICAL TRIAL: NCT02197780
Title: Calprotectin or Calgranulin C-test Before Undergoing Endoscopy: a Prospective Diagnostic Accuracy Study Comparing Two Fecal Biomarkers for Pediatric IBD
Brief Title: Head-to-head Comparison of Two Fecal Biomarkers to Screen Children for IBD
Acronym: CACATU
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Cisbio Bioassays (Industry)
Responsible Party: Principal Investigator, P.F. van Rheenen, Pediatric Gastroenterologist, University Medical Center Groningen
Other Study IDs: UMCG-2013N636
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Abdominal Pain; Rectal Bloodloss; Diarrhea; Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Irritable Bowel Syndrome
Keywords: Diagnostic accuracy; Fecal biomarker; Clinical Decision Rule; Cohort Study
MeSH Terms: conditions — Abdominal Pain; Diarrhea; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE:

A substantial proportion of children and teenagers with suspected inflammatory bowel disease (IBD) referred for endoscopy do not have the disease. The investigators designed a clinical decision rule that included a calprotectin stool test to discern which patients require further investigations. The accuracy of this diagnostic strategy is 88.5% with a low risk of missing IBD cases. Although the number of negative endoscopies was reduced after introduction of this strategy, still 22% of the referred children and teenagers underwent an unnecessary invasive test. S100A12 (calgranulin C) is a cytoplasmic protein secreted exclusively by activated neutrophils and this stool marker may be more IBD-specific than calprotectin.

OBJECTIVE:

To determine whether the specificity of S100A12 is superior to the specificity of calprotectin without sacrificing sensitivity

HYPOTHESIS:

Inclusion of the calgranulin C stool test will improve the specificity of the screening-strategy.

DETAILED DESCRIPTION:
DESIGN:

A prospective diagnostic accuracy study in several outpatient clinics for general paediatrics and several tertiary care hospitals in the Netherlands and Belgium.

STUDY POPULATION:

Eligible for inclusion are consecutive children and teenagers between 6 and 18 years who consult their pediatrician and have gastro-intestinal symptoms suggestive of IBD.

INTERVENTION:

Patients will be managed according to a calprotectin-based-referral strategy. Those with an elevated calprotectin level without colon pathogens are considered to have a high probability of IBD and may require referral for endoscopy (the preferred reference standard). Patients with confirmed gastrointestinal infection are advised to have their stools retested. Patients with normal calprotectin levels are considered to have a low probability of IBD and will therefore have a low change to be subjected to endoscopy. In these patients with low probablity of IBD an alternative reference standard may be performed, being clinical follow-up for 6 months. The decision for endoscopy or clinical follow up is up to the clinician's discretion, based on the combination of all symptoms, physical examination, blood results, fecal markers and colon pathogens.

Next to calprotectin, also S100A12 will be measured in all stool samples. We will perform a post hoc scenario analysis to compare the test characteristics of both fecal markers.

OUTCOME MEASURES:

The primary outcome measure is the difference in specificity between FC and S100A12 among the total number of non-IBD patients.

We adjusted our previously formulated outcome measure, being the proportion of patients with non-inflammatory conditions among the total number of patient subjected to endoscopy, for two reasons.

1. During an interim analysis in August 2016 the proportion of patients subjected to endoscopy was lower as expected (34% instead 46%). To reach the required amount of patients with the reference standard (endoscopy) we needed to extend the study for several months.
2. Triggered by a recently published paper by Naaktgeboren et al in the BMJ, we realized that our initial design would lead to biased results.

Secondary endpoints are the difference in sensitivity among the total number of patients with IBD and the diagnostic accuracy characteristics (sensitivity, specificity, positive predictive value, negative predictive value, area under the curve, best cut-off point) for both markers individually. All diagnostic accuracy characteristics will be calculated with 1) a pre-specified cut-off value based on literature, 2) the best cut-off point calculated with the data from this trial.

POWER/DATA ANALYSIS:

At the start of our trial we defined a sample size calculation, based on the previously described outcome measure including only patients with endoscopy. Based on a previous cohort study we expected that 46% of the recruited patients would undergo endoscopy. Using a sample size calculation based on independent samples calculated with a Fisher's exact test, we calculated that with 154 patients subjected to endoscopy the study would have 80% power to detect a 50% relative reduction of the primary outcome from 22% false positives with FC to 11% false positives with S100A12, at a one-sided alpha level of 0.05. The total number of patients to be recruited for this diagnostic accuracy study was therefore calculated at 335.

In the slipstream of the adjustment of the primary outcome measure, we adjusted our sample size. We now use McNemar's test for paired samples to compare the proportion of concordant and discordant results between FC and S100A12 in all patients with the disease or without the disease.

To calculate the new sample size we used a specificity of FC of 0.70, based on recent individual patient data meta-analysis of Degraeuwe and we expected S100A12 would lead to 50% relative improvement. A sample size of 130 subjects achieves 80% power to detect a difference of 0,15 between the two diagnostic tests whose specificities are 0,70 and 0,85. This procedure uses a two-sided McNemar test with a significance level of 0,05. The prevalence of non-IBD in the population is 0,64. The proportion of discordant pairs is 0,23.

ETHICAL CONSIDERATIONS:

The Medical Ethical Committee of the University Medical Center in Groningen has granted exemption from WMO-approval, as it involves the collection of data generated by routine medical care. After measurement of calprotectin levels and testing for microbial gut pathogens the residual material will be used for the measurement of calgranulin C levels. When patients and their parents give permission, residual feces will be stored for a maximum period of 15 years for future diagnostic research.

TIME SCHEDULE:

Total running time is 30 months, including 6 months to complete the follow up and 2 months for analysis and reporting.

ELIGIBILITY:
Eligible patients are those aged between 6 and 18 years with at least one of the following criteria:

* Persistent diarrhea (at least 4 wks)
* Recurrent abdominal pain with diarrhea (at least 2 episodes in 6 months)
* Rectal bloodloss
* Peri-anal disease

OR at least two of the following criteria:

* Involuntary weight loss
* First degree family member with IBD
* Anemia (HB < -2 SD for age and gender)
* Increased marker of inflammation (ESR >20 mm/hour or CRP >10 mg/L)
* Extra-intestinal symptoms (erythema nodosum, arthritis, uveitis, thromboembolism, aphtous ulcera)

We did not define any exclusion criteria.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible for inclusion are consecutive children and teenagers who consult their pediatrician and have gastro-intestinal symptoms suggestive of IBD. Participating centers are located in the Northern and Southern region of the Netherlands and the Flemish-speaking region of Belgium.
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The difference in specificity between FC and S100A12 among the total number of non-IBD patients. | 6 months

SECONDARY OUTCOMES:
The difference in sensitivity between FC and S100A12 among the total number of IBD patients. | 6 months
Diagnostic test accuracy characteristics for both FC and S100A12 | 6 months
  Calculate sensitivity, specificity, positive predictive value, negative predictive value, area under ROC-curve, best cut-off point. The sensitivity, specificity, positive predictive value and negative predictive value will be presented with 1) a pre-specified cutoff value based on literature and 2) with the best cut-off points from this trial

OTHER OUTCOMES:
Scenario analysis with the test accuracy for a combination of FC and S100A12 in (sub)selection of patients. | 6 months
  Scenario analysis with presentation of the number of true- and false positives and true- and false negatives for 1) only FC screening, 2) only S100A12 screening, 3) combination of FC and S100A12 screening, 4) combination of FC and S100A12 in sub-selection of patients with indeterminate result.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick F van Rheenen, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (19):
- Belgium (3):
  - Sint Vincentiusziekenhuis, Antwerp
  - University Hospital Antwerpen, Antwerp
  - University Hospital Gent, Ghent
- Netherlands (16):
  - ZGT Almelo, Almelo
  - Wilhelmina Ziekenhuis, Assen
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Nij Smellinghe, Drachten
  - Scheper Ziekenhuis, Emmen
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter ziekenhuis, Goes
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Tjongerschans, Heerenveen
  - Bethesda Hospital, Hoogeveen
  - Medisch Centrum Leeuwarden (MCL), Leeuwarden
  - Bravis ziekenhuis, Roosendaal
  - Refaja Ziekenhuis, Stadskanaal
  - Ommelander Ziekenhuis Groep, Winschoten
  - Isala Kliniek, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Van de Vijver E, Heida A, Ioannou S, Van Biervliet S, Hummel T, Yuksel Z, Gonera-de Jong G, Schulenberg R, Muller Kobold A, Verkade HJ, van Rheenen PF; CACATU CONSORTIUM. Test Strategies to Predict Inflammatory Bowel Disease Among Children With Nonbloody Diarrhea. Pediatrics. 2020 Aug;146(2):e20192235. doi: 10.1542/peds.2019-2235. Epub 2020 Jul 21. PMID 32694147
- [Derived] Heida A, Van de Vijver E, van Ravenzwaaij D, Van Biervliet S, Hummel TZ, Yuksel Z, Gonera-de Jong G, Schulenberg R, Muller Kobold A, van Rheenen PF; CACATU consortium. Predicting inflammatory bowel disease in children with abdominal pain and diarrhoea: calgranulin-C versus calprotectin stool tests. Arch Dis Child. 2018 Jun;103(6):565-571. doi: 10.1136/archdischild-2017-314081. Epub 2018 Mar 7. PMID 29514815
- [Derived] Heida A, Van de Vijver E, Muller Kobold A, van Rheenen P. Selecting children with suspected inflammatory bowel disease for endoscopy with the calgranulin C or calprotectin stool test: protocol of the CACATU study. BMJ Open. 2017 May 29;7(5):e015636. doi: 10.1136/bmjopen-2016-015636. PMID 28554936
- [Derived] Heida A, Dijkstra A, Dantuma SK, van Rheenen PF. A Cross-Sectional Study on the Perceptions and Practices of Teenagers With Inflammatory Bowel Disease About Repeated Stool Sampling. J Adolesc Health. 2016 Oct;59(4):479-81. doi: 10.1016/j.jadohealth.2016.06.009. Epub 2016 Aug 6. PMID 27506279